CLINICAL TRIAL: NCT00882531
Title: Evaluation of the Efficacy of Isotretinoin Versus Placebo in Terms of Response Rate Among Patients Presenting Papular-pustular Rosacea Resistant to Standard Therapy
Brief Title: Isotretinoin in Papular-Pustular Rosacea
Acronym: ISOROS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Bailleul-Biorga (Industry)
Collaborators: Quanta Medical (Industry)
Responsible Party: Clara Jaramillo, laboratoires BAILLEUL BIORGA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISOROS
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Papular-pustular Rosacea
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isotretinoin (Experimental)
  Interventions: Drug: isotretinoin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: isotretinoin — 0.25 mg/kg, 1 per day, 4 month of treatment
  Arms: Isotretinoin
Drug: placebo
  Arms: placebo

SUMMARY:
A national, multicentre, prospective, randomised, double-blind, phase III study in 2 parallel groups of isotretinoin versus placebo in patients presenting papular-pustular rosacea resistant to standard therapy. A non-balanced group (2 isotretinoin /1 placebo) design was selected since, given the nature of the study disease, fewer patients will receive the placebo than active isotretinoin.

Treatment duration for each patient : 4 months, with monthly evaluation Follow-up at 2 months and 4 months for patients responsive after 4 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patients presenting papular-pustular rosacea (characterised by at least 8 lesions (papules and/or pustules)
* resistant for at least 3 months in the last two years to standard treatment comprising systemic antibiotics (cyclins) with or without topical therapy
* Full compliance with a two-week wash-out period for all other topical and systemic treatments for rosacea at the time of selection
* For women of childbearing age, use of a minimum of one "effective" contraceptive method for at least one month and willingness to continue using an effective contraceptive method continuously throughout the study duration and for at least one month after the end of treatment.
* Women of childbearing age must provide consent for pregnancy testing before the start of treatment, monthly throughout treatment and 5 weeks after the end of treatment.
* Negative pregnancy test results from within the last 3 days (for female subjects of childbearing age)
* No laboratory abnormalities in standard tests
* Social Security medical cover
* Provision of written and dated informed consent to take part in the study

Exclusion Criteria:

* Patients already receiving isotretinoin for rosacea or within the last 12 months for acne
* Patients presenting perioral dermatitis
* Patients presenting miliary lupoid
* Patients presenting cortisone-induced rosacea
* Pregnant or breast-feeding women
* Patients with repeated and habitual heavy physical activity
* Patients with known hepatic impairment presenting cytolysis as attested by laboratory results
* Patients presenting hyperaemia
* Patient presenting hypervitaminosis A
* Patients with a history of hypersensitivity to isotretinoin
* Patients with allergy to soy oil
* Patients on tetracycline
* Patients with depression treated at the time of selection
* Patients currently taking part in having taken part in another study in the last 3 months prior to inclusion in the present study
* Patients protected by law (under guardianship or trusteeship)
* Patients unable to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine numbers of patients responding to treatment for 4 months with isotretinoin (patients were considered as responders if their number of papular-pustular lesions fell by at least 90% after 4 months of treatment)

SECONDARY OUTCOMES:
Improvement in patients' quality of life using the reduced Skindex-France QoL scale (30 items)
Change in severity of other symptoms of rosacea (burning sensation, erythema, telangiectasia, vasomotor flush, etc)
Patient satisfaction (on a visual analogue scale)
Global treatment efficacy (global assessment)
Relapse rates at 8 months (after start of treatment)
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSIDOW, Professor, Principal Investigator